CLINICAL TRIAL: NCT04599361
Title: Health Care Analysis on Myocardial Revascularization in Patients With Chronic Coronary Heart Disease (CHD)
Acronym: REVASK
Status: Completed | Type: Observational
Sponsor: InGef - Institute for Applied Health Research Berlin GmbH (Industry)
Collaborators: University of Education Freiburg (Unknown); Deutsche Gesellschaft für Thorax-, Herz- und Gefäßchirurgie (DGTHG) (Unknown); Stiftung Institut fuer Herzinfarktforschung (Other); Universitätsklinikum Köln (Other); BARMER (Other); Techniker Krankenkasse (Other)
Responsible Party: Sponsor
Other Study IDs: 01VSF18010; DRKS00022175 (Registry Identifier: German clinical trials register)
Record Dates: First submitted 2020-09-11; First posted 2020-10-22 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Coronary Heart Disease
Keywords: Chronic coronary heart disease; myocardial revascularization; heart team; decision making; cardiology; heart surgery
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with CHD: outpatient cardiology practices, hospitals with a cardiology department and hospitals with a cardiology and heart surgery department (n=20) in Germany Patients with chronic coronary heart disease and 2- or 3-vessel or main-vessel disease who are being treated at one of the recruitment sites with a promptly planned intervention for myocardial revascularization who are insured with pre-specified German health insurance companies (BARMER or TK)
  Patients will receive questionnaires.

SUMMARY:
Myocardial infarction and chronic coronary heart disease (cCHD) are the most frequent causes of death in Germany. Treatment options include widening of the narrowed / blocked coronary vessel via catheter and stent or bypass surgery in which the narrowed vessel sites are bridged. The "German National Disease Management Guideline on cCHD" helps doctors to decide which treatment is most appropriate for the severity of vascular damage and possible concomitant diseases of the patient. Nevertheless, there are other factors determining treatment decision. For example, the equipment or preferences of the hospital or department in which patients are admitted, play a role in the decision.

The aim of the REVASK project is to investigate whether and to what extent the collaboration of cardiology and heart surgery specialists in so-called "heart teams" influences the decision on therapy.

For this purpose, doctors and patients will be interviewed about how the treatment decision was made and how satisfied both sides are with the outcome of the treatment and the decision. In addition, claims data from several German health insurance companies (Techniker, BARMER, Betriebs- und Innungskrankenkassen) will be analyzed. Treatment data, which is documented as usual by the treating medical staff and passed on to the health insurance companies for accounting purposes, is used. Furthermore, treatment data recorded in the registers of the professional societies is analyzed.

ELIGIBILITY:
Inclusion Criteria:

* with chronic coronary heart disease
* and 2- or 3-vessel or main-vessel disease
* who are being treated at one of the recruitment sites
* with a promptly planned intervention for myocardial revascularization
* who are insured with pre-specified German health insurance companies (BARMER or TK)

Exclusion Criteria:

-

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: outpatient cardiology practices, hospitals with a cardiology department and hospitals with a cardiology and heart surgery department (n=20) in Germany
Sampling Method: Non-Probability Sample
Enrollment: 385 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Guideline compliance | 2 years
  Guidelines-compliant therapy in patients with chronic CHD (2- or 3-vessel or main vessel disease) according to German National Disease Management Guideline on chronic coronary heart disease

SECONDARY OUTCOMES:
Heart teams | 2 years
  Frequency and quality of heart teams
Patient participation | 2 years
  extent of patient participation in the decision making process
Decision making process | 2 years
  importance of clinical parameters in the decision-making process (e.g. syntax scores, iFR, FFR)

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Walker, Dr. med., Study Chair — InGef - Institute for Applied Health Research Berlin GmbH; Spittelmarkt 12, 10117 Berlin; Andreas Beckmann, Dr. med., Principal Investigator — Deutsche Gesellschaft für Thorax-, Herz- und Gefäßchirurgie (DGTHG); Uwe Zeymer, Prof. Dr. med., Principal Investigator — Stiftung Institut für Herzinfarktforschung (IHF); Peter Ihle, Principal Investigator — PMV forschungsgruppe, Universitätsklinikum Köln; Ursula Marschall, Dr.med., Principal Investigator — BARMER; Ines Meier, Dr., Principal Investigator — Techniker Krankenkasse
Locations (1):
- Pädagogische Hochschule Freiburg Public Health & Health Education, Freiburg im Breisgau, Germany

IPD SHARING:
Plan to Share IPD: Yes
Research data can be shared with persons or institutions with a legitimate scientific interest after consultation in the consortium and only in pseudonymised form and within the scope of the EU-GDPR

REFERENCES:
- See also: The official website of the REVASK project — https://revask.de/